CLINICAL TRIAL: NCT07225374
Title: A Prospective Phase II Study of Adjuvant Cisplatin-Based Chemotherapy Followed by Maintenance Avelumab in Upper Tract Urothelial Carcinoma
Brief Title: Cisplatin-Based Chemotherapy Followed by Maintenance Avelumab in UTUC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park, Se-Hoon, Samsung Medical Center, Principal Investigator, Clinical Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-03-132; KCT0010668 (Other: CRIS)
Record Dates: First submitted 2025-09-16; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Upper Tract Urothelial Carcinoma
MeSH Terms: interventions — avelumab; Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Avelumab) (Experimental): It is a single arm study and in this arm patients who meet all of the inclusion criteria and none of the exclusion criteria will receive avelumab 10 mg/kg as a
  1-h infusion every 2 weeks. Avelumab will repeat every 2 weeks on an outpatient basis and continued until disease recurrence, unacceptable toxicity, consent withdrawal, or for a maximum of 1 year.
  Interventions: Drug: Avelumab 10 mg/kg; Procedure: Screening; Procedure: Best Supportive Care (BSC); Other: Follow-up plan

INTERVENTIONS:
Drug: Avelumab 10 mg/kg — Patients who meet all of the inclusion criteria and none of the exclusion criteria will receive avelumab 10 mg/kg as a
  1-h infusion every 2 weeks. Avelumab will repeat every 2 weeks on an outpatient basis and continued until disease recurrence, unacceptable toxicity, consent withdrawal, or for a maximum of 1 year.
Procedure: Screening — Screening numbers are endowed to all patients who sign the informed consent forms.
  These screening numbers are used as 'Subject Identification Code" along with patient initials. Patients withdrawn from the study retain their screening number. New patients must always be allotted with a new screening number.
Procedure: Best Supportive Care (BSC) — All study subjects will be also eligible to receive best supportive care (BSC) defined as any standard supportive measures that are not considered a primary treatment of the disease under study, including the use of growth factors (i.e. G-CSF) for myelosuppression, analgesics and transfusion of blood products. BSC will be provided at the discretion of the investigators.
Other: Follow-up plan — All patients are to have a clinic visit every 2 weeks (+3 days) during during study treatment. Tumor assessments will be performed at screening and approximately every 12 weeks, or sooner if deemed necessary by the investigator. A tumor assessment will be performed upon treatment discontinuation (End of Treatment visit) if the reason for discontinuation is other than disease progression and no tumor assessment was performed in the prior 12 weeks, or a tumor assessment is required for the confirmation of DFS.

SUMMARY:
A Prospective Phase II Study of Adjuvant Cisplatin-Based Chemotherapy followed by Maintenance Avelumab in Upper Tract Urothelial Carcinoma

DETAILED DESCRIPTION:
Upper tract urothelial carcinoma (UTUC), including those that arise in the renal pelvis or in ureter, are relatively uncommon but highlyinvasive. Although radical surgery followed by adjuvant chemotherapy is considered a standard in the management of UTUC, a significant percentage of patients experience recurrence, leading to a poor prognosis. Nivolumab has been investigated for adjuvant treatment in the other trial, but unfortunately, a better DFS was not observed in patients with UTUC. Given the promising efficacy of the maintenance avelumab following first-line chemotherapy, the maintenance strategy looks promising in the adjuvant setting of curatively-resected UTUC.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 19 years or more
* Must have histologically or cytologically proven UTUC arising from renal pelvis and/or ureter.
* Must have histological evidence of high-risk muscle-invasive disease (i.e., pT2~ T4) and/or N+ disease.
* Must have an ECOG performance status of 0 to 1
* Received at least 3 or 4 cycles of adjuvant cisplatin-based chemotherapy, and proved to have no evidence of disease recurrence with imaging studies, urine cytology and cystoscopy
* At least 3 weeks since the last surgical procedures or chemotherapy prior to enrolment. Subjects must have recovered to <Grade 2 from all acute toxicities or toxicity must be deemed irreversible by the investigator.
* Adequate marrow function without growth factor support or transfusion dependency A. Neutrophil 1,500 cells/μL or more B. Platelet count 100,000/μL or more C. Hemoglobin 9.0 g/dL or more
* Adequate renal function with serum creatinine 1.5 x ULN or a calculated creatinine clearance ≥ 50 mL/min using the CockcroftGault or MDRD formulas
* Adequate hepatic function A. Bilirubin 1.5 times upper limit of normal (x ULN) or less; does not apply to subjects with Gilbert's syndrome diagnosed as per institutional guidelines. B. AST (SGOT) and ALT (SGPT) 3 x ULN or less; if liver metastases are present, then 5 x ULN is allowed.
* Women of childbearing potential must use effective contraception continuously for at least 30 days after the final dose of avelumab. At least one method classified as "highly effective" (failure rate < 1%) must be employed (see Table 1).
* Written and voluntary informed consent understood, signed and dated.
* Negative serum or urine pregnancy test at screening for women of childbearing potential.

Exclusion Criteria

* Ongoing treatment with an anticancer agent not contemplated in this protocol
* Radiologic finding consistent with metastatic disease
* Severe medical or psychological illness that preclude participation to study, including any history of clinically relevant coronary artery disease or myocardial infarction within the last 3 years, New York Heart Association (NYHA) grade III or greater congestive heart failure, cerebrovascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation
* Non-tolerable > Grade 2 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1
* Major surgery, other than diagnostic surgery or transurethral resection, within 4 weeks prior to Cycle 1 Day 1, without complete recovery
* Double primary cancer of other site(s) or a history of other malignancies, except for cured ones at the discretion of investigator
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Subjects who have exhibited allergic reactions to study treatment.
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
* Subject with legal incapacity or limited legal capacity. Dementia or significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication). 12) Active autoimmune disease requiring systemic immunosuppressive treatment. Patients with controlled autoimmune disease not requiring systemic immunosuppressive treatment including diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
* Persisting toxicity related to prior therapy (NCI CTCAE Grade >

  1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Lactating Women Must discontinue breastfeeding during study treatment and for at least 30 days after administration of the final dose of study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2029-07-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | In brief, CT scans (or MRIs) will be performed every 12 weeks during study treatment, through study completion, until progression of disease or 1 year starting from enrollment of study.
  Disease-free survival (DFS)

SECONDARY OUTCOMES:
Progression free survival | All subjects will be evaluated PFS as the time from the date of first study treatment to the date of disease progression or death, whichever comes first through the study, or 1 year starting from enrollment of study.
  Progression will be evaluated in this study using the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: SE HOON PARK, MD,PhD, Principal Investigator — SamsungMedicalCenter
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: Yes